CLINICAL TRIAL: NCT06008327
Title: Comparison Of The Outcome Of Treatment Of Topical 15% Trichloroacetic Acid Versus Topical 0.05% Tretinoin In The Treatment Of Acanthosis Nigricans
Brief Title: Comparison Of Outcome Of Treatment OF Topical 15%TCA VS Topical 0.05% Tretinoin In Treatment Of Acanthosis Nigricans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Dr Khadijah, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.F2-81/2022-GENL/254/JPMC
Record Dates: First submitted 2023-03-22; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Acanthosis Nigricans
MeSH Terms: conditions — Acanthosis Nigricans | interventions — Trichloroacetic Acid; Tretinoin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Topical 15% Trichloroacetic acid (Experimental): 15 % Trichloroacetic acid (TCA) and 0.05%Tretinoin for 02 months Trichloroacetic acid, a superficial chemical exfoliative agent has shown efficacy in treating acanthosis nigricans. 9-10 Data from this would help in establishing it as a treatment of choice thereby lead to reduction in cost and benefit the patient both financially and psychologically.
  Interventions: Drug: Topical 15% Trichloroacetic acid
- Group B Topical 0.05% Tretinoin (Experimental): Topical tretinoin is the first choice of drug in the treatment of acanthosis nigricans. Despite several therapeutic modalities, acanthosis nigricans (AN) remains a difficult dermatosis to treat.
  Interventions: Drug: Topical 15% Trichloroacetic acid

INTERVENTIONS:
Drug: Topical 15% Trichloroacetic acid — Recently trichloroacetic acid (TCA), a superficial chemical exfoliative agent has shown efficacy in treating acanthosis nigricans. Data from this would help in establishing it as a treatment of choice thereby lead to reduction in cost and benefit the patient both financially and psychologically.
  Other Names: Topical 0.05% Tretinoin

SUMMARY:
Acanthosis nigricans (AN) is a dermatosis with aesthetic implications and is characterized by the focal or diffuse development of a velvety, hyperpigmented cutaneous thickening in intertriginous areas. Trichloroacetic acid (TCA), a superficial chemical exfoliative agent has shown efficacy in treating acanthosis nigricans. Data from this would help in establishing it as a treatment of choice thereby lead to reduction in cost and benefit the patient both financially and psychologically.

DETAILED DESCRIPTION:
Acanthosis nigricans is common, although exact prevalence depends upon the racial makeup of the population studied. Exact pathogenesis is unknown, elevated insulin concentrations result in direct and indirect activation of IGF-1 receptors on keratinocytes and fibroblasts, leading to proliferation. This hyperpigmentation, which has poorly defined borders, usually occurs in skin fold areas symmetrically, such as the back of the neck, axilla and groin, and may rarely involve oral mucosa. The lesions may be related to a wide range of benign conditions and may occur as a paraneoplastic manifestation of various potentially fatal malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will present with acanthosis nigricans as per operational definition will be included in the study.

  * Either gender.
  * Age 20-50 years.

Exclusion Criteria:

Pregnancy.

* Breastfeeding.
* Patients with history of skin resurfacing by dermabrasion, chemical peels and facial laser within the preceding 9 months.
* Patients with history of hypersensitivity.
* Malignant Acanthosis Nigricans.
* Drug Induced Acanthosis Nigricans.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
EFFICACY OF TOPICAL 15%TRICHLOROACETIC ACID VERSUS 0.05% TOPICAL TRETINOIN IN ACANTHOSIS NIGRICANS | It will be assessed upto 02 months
  Efficacy will be assessed by taking serials photographs before and after treatment shown efficacy in treating acanthosis nigricans. Data from this would help in establishing it as a treatment of choice thereby lead to reduction in cost and benefit the patient both financially and psychologically.

CONTACTS AND LOCATIONS:
Overall Officials: Parisa Sanawar, FCPS, Principal Investigator — Jpmc; Nazia Jabeen, FCPS, Principal Investigator — Jpmc; Fazia Inam, FCPS, Principal Investigator — Jpmc
Locations (1):
- JPMC, Karachi, Sindh, Pakistan